CLINICAL TRIAL: NCT04522947
Title: Modifiable Predictors of Neural Vulnerabilities for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other); University of Utah (Other); Gretchen Swanson Center for Nutrition (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20317; R01DK125651 (NIH)
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All participants complete the same fMRI protocol which includes delivery of appetizing taste stimuli and tasteless stimuli while in the scanner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI (Experimental): Participants are delivered sips of appetizing tastes (milkshake) and tasteless solution throughout the task while in the MRI scanner.
  Interventions: Other: Milkshake fMRI

INTERVENTIONS:
Other: Milkshake fMRI — While in the MRI scanner, the participant is shown a cue indicating the impending delivery of either milkshake or tasteless solution, followed by a brief blank screen, then delivery of the sip, and then a swallow cue. This procedure is repeated throughout the task.

SUMMARY:
The purpose of this study is to examine patterns of neural activation in a priori selected brain regions associated with reward process during anticipation and delivery of appetizing food stimuli (milkshake sips) among young adults.

DETAILED DESCRIPTION:
This observational trial seeks to examine neural activation patterns in a food reward sensitivity task. The study uses the "milkshake" MRI task to assess individual food reward sensitivity in a sample of young adult participants. Participants are presented with a series of trials in which a visual cue is provided (either a glass of milkshake or water), followed by delivery of a sip of the corresponding liquid. Activation in a priori regions associated with reward processing is measured via blood oxygen level-dependent (BOLD) signal, both in response to the cue and actual delivery of the sip. Explicating patterns of reward processing for appetizing food stimuli holds potential to inform understanding of the neural underpinnings of obesity risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Previous participation in the Preschool Problem Solving Study OR lived in Lancaster County, NE for at least part of high school

Exclusion Criteria:

* Contraindications for functional magnetic resonance imaging (fMRI):
* metal in body
* pregnancy
* braces
* non-removal piercings
* hair extensions
* As of 8/13/21, for individuals who were not in the Preschool Problem Solving Study but are invited to participate in the current study because they lived in Lancaster County for at least part of high school, the maximum age for eligibility is 20 years of age.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Nelson, Ph.D., Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

RESULTS

PARTICIPANT FLOW:
Groups:
- fMRI Milkshake Task: Participants are delivered sips of appetizing tastes (milkshake) and tasteless solution throughout the task while in the MRI scanner.
  Milkshake fMRI: While in the MRI scanner, the participant is shown a cue indicating the impending delivery of either milkshake or tasteless solution, followed by a brief blank screen, then delivery of the sip, and then a swallow cue. This procedure is repeated throughout the task.
Period: Overall Study
Arm/Group | fMRI Milkshake Task
Started | 187
Completed | 187
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | fMRI Milkshake Task
Number analyzed (Participants) | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 187
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 162
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 133
  More than one race | 24
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 187

OUTCOME MEASURES:

1. Primary Outcome: Caudate Activation for Sip Cue
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the caudate for all milkshake cue trials versus all tasteless solution cue trials (milkshake>tasteless) after receiving the cue but before the delivery of the actual sip.
Time Frame: 7 seconds after cue is presented
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | -0.026264341 (0.261413915)

2. Primary Outcome: Putamen Activation for Sip Cue
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the putamen for all milkshake cue trials versus all tasteless solution cue trials (milkshake>tasteless) after receiving the cue but before the delivery of the actual sip.
Time Frame: 7 seconds after cue is presented
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | -0.020653429 (0.23259893)

3. Primary Outcome: Insula Activation for Sip Cue
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the insula for all milkshake cue trials versus all tasteless solution cue trials (milkshake>tasteless) after receiving the cue but before the delivery of the actual sip.
Time Frame: 7 seconds after cue is presented
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | -0.058804599 (0.1660244)

4. Primary Outcome: Caudate Activation for Sip Delivery
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the caudate for all milkshake trials versus all tasteless solution trials (milkshake>tasteless) upon delivery of the actual sip.
Time Frame: 7 seconds after delivery of sip
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | -0.01520067 (0.269324341)

5. Primary Outcome: Putamen Activation for Sip Delivery
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the putamen for all milkshake trials versus all tasteless solution trials (milkshake>tasteless) upon delivery of the actual sip.
Time Frame: 7 seconds after delivery of sip
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | -0.010750489 (0.211345119)

6. Primary Outcome: Insula Activation for Sip Delivery
Description: MRI blood oxygen level-dependent (BOLD) activity signal in the insula for all milkshake trials versus all tasteless solution trials (milkshake>tasteless) upon delivery of the actual sip.
Time Frame: 7 seconds after delivery of sip
Measure: Mean (Standard Deviation); unit: activation beta value
Arm/Group | fMRI
Number analyzed (Participants) | 187
activation beta value | 0.084583225 (0.173758221)

ADVERSE EVENTS:
Time Frame: During the session in which the milkshake task trial was conducted
Arm/Group | fMRI Milkshake Task
All-Cause Mortality (participants affected / at risk) | 0/187
Serious Adverse Events (participants affected / at risk) | 0/187
Other Adverse Events (participants affected / at risk) | 0/187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04522947/Prot_SAP_001.pdf
  • Informed Consent Form (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT04522947/ICF_000.pdf